CLINICAL TRIAL: NCT06686940
Title: Photoplethysmography (PPG) Algorithm With Smartwatch in Evaluation of Atrial Fibrillation Burden
Acronym: Polaris-AF
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2024100; KS2024100 (Other: Chengdu Xinjikang Technology Co., Ltd)
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation burden; Photoplethysmography; Wearable devices.
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Photoplethysmography data、Electrocardiogram data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intervention group — The monitoring effect of a smart electrocardiogram watch based on the PPG algorithm on atrial fibrillation burden.

SUMMARY:
The purpose of this study is to evaluate the monitoring effect of a smart electrocardiogram watch based on the PPG algorithm on atrial fibrillation burden.

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation patients diagnosed by electrocardiogram
2. Willing to use long-range electrocardiogram monitoring equipment

Exclusion Criteria:

1.Patients who are allergic to electronic devices or unable to wear watches

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with atrial fibrillation who meet age and health criteria can use electrocardiographic watches for long-term monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2034-12-30 (Estimated); Study Completion 2034-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | December 30, 2024 to Decemberr 30, 2034
  all-cause death, cardiovascular death, myocardial infarction, heart failure, stroke, peripheral vascular disease, recurrence of atrial fibrillation diagnosed by electrocardiogram, palpitations symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No